CLINICAL TRIAL: NCT01406015
Title: Mineralocorticoid Receptor and Obesity Induced Cardiovascular Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rajesh K. Garg, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2009P-000311
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin resistance; Mineralocorticoid receptor
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Active Comparator)
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 50 mg once daily for 6 weeks.
  Arms: Spironolactone
Drug: Placebo — Placebo-matching spironolactone once daily for 6 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if spironolactone, a drug that blocks the action of aldosterone, can make the blood vessels work better in people with obesity. The investigators also want to find out whether spironolactone causes changes in levels of insulin and markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Good health as evidenced by history and physical exam
3. Body Mass Index (BMI): >30 kg/m2 and <45 kg/m2

Exclusion criteria:

1. Medical illnesses other than treated hypothyroidism
2. Blood Pressure (BP) >135/85 or systolic BP <90 mm Hg
3. Hepatic disease (transaminase > 3 times normal)
4. Renal impairment (Creatinine clearance <60 ml/min)
5. Baseline serum Potassium (K) >5.0 mmol/L
6. History of drug or alcohol abuse
7. Allergies to spironolactone
8. Participation in any other concurrent clinical trial
9. Women using oral contraceptives within the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brown JM, Williams JS, Luther JM, Garg R, Garza AE, Pojoga LH, Ruan DT, Williams GH, Adler GK, Vaidya A. Human interventions to characterize novel relationships between the renin-angiotensin-aldosterone system and parathyroid hormone. Hypertension. 2014 Feb;63(2):273-80. doi: 10.1161/HYPERTENSIONAHA.113.01910. Epub 2013 Nov 4. PMID 24191286
- [Derived] Garg R, Kneen L, Williams GH, Adler GK. Effect of mineralocorticoid receptor antagonist on insulin resistance and endothelial function in obese subjects. Diabetes Obes Metab. 2014 Mar;16(3):268-72. doi: 10.1111/dom.12224. Epub 2013 Oct 31. PMID 24125483

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone: Spironolactone 50 mg once daily for 6 weeks.
Period: Overall Study
Arm/Group | Spironolactone | Placebo
Started | 19 | 19
Completed | 16 | 16
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on the total number of participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11.6) | 40 (12.3) | 43.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 6 | 4 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 38 (6.6) | 36 (4.6) | 36.8 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-ischemic Dilatation
Description: Ultrasonography of the brachial artery was performed to evaluate endothelial function by flow mediated dilatation (FMD) studies. A blood pressure cuff was placed on the participant's upper arm and was compressed for 5 minutes. After release of compression, brachial artery diameter and blood flow velocity were measured. FMD was expressed as the percentage change in brachial artery diameter. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 6
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: percent dilalation
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 16 | 16
percent dilalation
  Baseline | 9.6 (7.8) | 10.2 (6.9)
  Change from Baseline at Week 6 | -1.2 (6.1) | -2.0 (4.7)

2. Secondary Outcome: Change From Baseline in Para-aminohippurate (PAH) Clearance
Description: Renal plasma blood flow was determined by clearance of para-aminohippurate (PAH). A loading dose of PAH (8 mg/kg) was given intravenously followed by a 1 hour constant infusion of PAH at a rate of 12 mg/minute (min). Plasma samples were obtained at Baseline and at 50 and 60 minutes. PAH clearance was calculated from the plasma levels and infusion rates and reported in millimeters (mL)/minute (min). A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 6 (Prior to PAH infusion and at 50 and 60 minutes post PAH infusion)
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 16 | 16
mL/min
  Baseline | 488 (80) | 521 (116)
  Change from Baseline at Week 6 | -2.3 (28.7) | -5.2 (25.3)

3. Secondary Outcome: Change From Baseline in Markers of Inflammation
Description: Blood was to be collected and tested for Tumor Necrosis Factor Alpha (TNF-α) and Monocyte Chemotactic Protein-1 (MCP-1), markers of inflammation; However, due to lack of funding, blood samples were not analyzed and data for levels of inflammation markers were not collected.
Time Frame: Baseline and Week 6
Population: Analysis was not performed.
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Insulin Sensitivity Index (ISI)
Description: Insulin sensitivity was measured using the 75 gram (G) glucose tolerance test. Participants ingested 75 grams of glucose in 300-400 milliliters (mL) of water over 5 minutes. Blood samples were taken before ingesting glucose and then every 30 minutes for 120 minutes. Insulin sensitivity index was calculated by Matsuda and Defronzo's formula using the values obtained. A positive change from Baseline (increase in insulin sensitivity) indicates improvement.
Time Frame: Baseline and Week 6 (Prior to ingesting glucose and every 30 minutes for 120 minutes)
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: IS index
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 16 | 16
IS index
  Baseline | 3.7 (1.4) | 4.6 (3.7)
  Change from Baseline at Week 6 | -0.1 (0.8) | -1.1 (2.7)

5. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Insulin resistance was measured using the 75 G glucose tolerance test. Participants ingested 75 grams of glucose in 300-400 mL of water over 5 minutes. Blood samples were taken before ingesting glucose and then every 30 minutes for 120 minutes. HOMA-IR was calculated using the Insulin and glucose levels obtained. A negative change (decrease in insulin resistance) indicates improvement.
Time Frame: Baseline and Week 6 (Prior to ingesting glucose and every 30 minutes for 120 minutes)
Population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: IR index
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 16 | 16
IR index
  Baseline | 2.7 (1.2) | 3.4 (3.2)
  Change from Baseline at Week 6 | 0.1 (1.1) | 0.1 (4.4)

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Spironolactone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes